CLINICAL TRIAL: NCT00517946
Title: An Investigation to Evaluate the Technique of MRI as an Assessment of the Effect of Anti-allergy Drug Treatment on Internal Nasal and Sinus Mucosal Anatomy Following Intranasal Allergen Challenge in Subjects With Seasonal Allergic Rhinitis.
Brief Title: A Study To Investigate If MRI Scanning Is Effective At Seeing What Hayfever Drugs Do In Nasal Passage.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: RES101509
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Seasonal Allergic Rhinitis; Sinusitis
Keywords: anti-allergy.; seasonal allergic rhinitis (SAR),; intranasal allergen challenge,; MRI,
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Sinusitis | interventions — Pseudoephedrine; Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pseudoephedrine hydrochloride
Drug: cetirizine hydrochloride
  Other Names: pseudoephedrine hydrochloride

SUMMARY:
The purpose of this study is to establish whether MRI scanning is a sensitive measure of the effects of existing drug treatments on nasal dimensions following challenge with intranasal allergen in subjects with hayfever. If successful this technique could be applied to increase confidence for internal decision making and ultimately may be used to assess how effective a new drug treatment is.

ELIGIBILITY:
Inclusion Criteria:

* A medically diagnosed hay fever patient who is otherwise healthy.
* Aged 18 to 60 years.
* Body mass index less than 30 kg/m² with weight range of 50kg (females 45kg) to 100kg.
* A positive skin prick test (wheal = 3mm) for grass pollen at or within 12 months of starting the study and/or a positive RAST (= class 2) for grass pollen at or within 12 months of starting the study.
* Baseline FEV1 = 80% predicted and a baseline FEV1/FVC = 70% predicted (using standard predicted guidelines).
* Capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all study measurements.

Exclusion Criteria:

* Pregnant or nursing females.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception.
* On examination the subject is found to have any nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, or nasopharyngeal surgery.
* Recent (within 3 weeks) or ongoing chest infection which in the physician responsible opinion renders the subject unsuitable for participation in the study.
* The subject has a history or current evidence of perennial rhinitis, sinusitis, or any other condition potentially or directly involving the nasal cavity, sinuses or nasopharynx.
* A history of any medical condition that would not allow the use of pseudoephedrine (e.g. hypertension, diabetes mellitus, ischaemic heart disease, raised intraocular pressure, hyperthyroidism, benign prostatic hyperplasia) or cetirizine (eg. antihistamine hypersensitivity).
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge.
* The subject has a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject has participated in another study during the previous 3 months.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, oral contraceptives and herbal remedies.
* The subject regularly, or on average, drinks more than 4 units of alcohol per day - where 1 unit = ½ pint of beer (284mL), or 1 glass of wine (125mL), or 1 measure of spirit (25mL).
* The subject smokes more than 5 cigarettes per day.
* The subject has a history of porphyria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Cross-sectional airspace area (and thus also airspace volume) of the nasal passages | at 1hr post-dose and 30-60mins post-allergen challenge.

SECONDARY OUTCOMES:
Volume of fluid identified adjacent to the airspace. Mucosal surface area. Nasal cavity volume. Nasal tissue volume derived from the nasal cavity volume less airspace and fluid volumes. | At 1hr post-dose and 30-60mins post-allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom